CLINICAL TRIAL: NCT00783094
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Design Study to Evaluate the Efficacy and Safety of Tadalafil Once-a-Day Dosing for 12 Weeks Followed by an Open-Label Extension to Evaluate the Long-Term Safety and Efficacy of Tadalafil in Japanese Men With Signs and Symptoms of Benign Prostatic Hyperplasia
Brief Title: Study of Tadalafil Once-a-Day for 12 Weeks in Japanese Men With Benign Prostatic Hyperplasia Followed by an Open-Label Extension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12757; H6D-JE-LVIA (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Results first posted 2010-07-28 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tadalafil 2.5 milligrams (mg) (Experimental): 2.5 mg tadalafil tablet by mouth once a day for 12 weeks followed by 5 mg tadalafil tablet by mouth once a day for 42 weeks.
  Interventions: Drug: Tadalafil 2.5 mg
- Tadalafil 5 mg (Experimental): 5 mg tadalafil tablet by mouth once a day for 12 weeks then continue 5 mg tadalafil tablet by mouth once a day for 42 weeks.
  Interventions: Drug: Tadalafil 5 mg
- Placebo (Placebo Comparator): Placebo tablet taken by mouth once a day for 12 weeks.
  Then subjects may take 5 mg tadalafil tablet by mouth once a day for 42 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil 2.5 mg — oral, daily
  Other Names: LY450190; Cialis
  Arms: Tadalafil 2.5 milligrams (mg)
Drug: Tadalafil 5 mg — oral, daily
  Other Names: LY450190; Cialis
  Arms: Tadalafil 5 mg
Drug: Placebo — oral, daily
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, parallel-design to compare the efficacy and safety of tadalafil once-a-day dosing versus placebo for 12 weeks followed by an open-label extension to evaluate the long-term safety and efficacy of tadalafil in Japanese men with signs and symptoms of benign prostatic hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* Japanese Males, 45 years old or older, with benign prostatic hyperplasia (BPH) for at least 6 months prior to Visit 1 and an International Prostate Symptom Score (IPSS) greater than or equal to 13 at Visit 2.
* Agree not to use any other approved or experimental pharmacologic BPH, erectile dysfunction (ED), and/or overactive bladder (OAB) treatments at any time during the study.
* Have not taken Finasteride or Dutasteride therapy, Anti-androgenic hormone or any other BPH therapy, ED or OAB therapy for specified duration of time prior to Visit 2.

Exclusion Criteria:

* Prostate specific antigen (PSA) score beyond acceptable range defined for study at Visit 1.
* History of urinary retention or lower urinary tract (bladder) stones within 6 months of Visit 1.
* History of urethral obstruction due to stricture, valves, sclerosis, or tumor at Visit 1.
* Clinical evidence of prostate cancer at Visit 1.
* Clinical evidence of any of the bladder or urinary tract conditions, which may affect lower urinary tract symptom at Visit 1.
* History of cardiac conditions, including Angina requiring certain treatment with nitrates, unstable angina defined for study, positive cardiac stress test before starting the study.
* History of significant central nervous system (CNS) injuries (including stroke or spinal cord injury) within 6 months of Visit 1.
* Use of any nitrates, cancer chemotherapy, androgens, antiandrogens, estrogens, luteinizing hormone-releasing hormone (LHRH) agonists/antagonists, or anabolic steroids at Visit 1.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- Japan (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Tadalafil 2.5 mg: 2.5 milligrams (mg) tadalafil tablet by mouth once a day for 12 weeks followed by 5 mg tadalafil tablet by mouth once a day for 42 weeks.
Period: Randomized Double-Blind Treatment Period
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Started | 142 | 140 | 140
Completed | 135 | 128 | 131
Not Completed | 7 | 12 | 9
Not completed — Adverse Event | 4 | 5 | 5
Not completed — Lack of Efficacy | 0 | 2 | 1
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 2
Period: Open-Label Extension Period
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Started | 135 | 128 | 131
Completed | 113 | 109 | 101
Not Completed | 22 | 19 | 30
Not completed — Adverse Event | 12 | 7 | 16
Not completed — Death | 0 | 0 | 1
Not completed — Protocol Violation | 4 | 5 | 7
Not completed — Withdrawal by Subject | 1 | 1 | 3
Not completed — Physician Decision | 4 | 2 | 3
Not completed — Lack of Efficacy | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo | Total
Number analyzed (Participants) | 142 | 140 | 140 | 422
Age Continuous [Mean (Standard Deviation); unit: years] | 66.4 (7.4) | 66.9 (7.7) | 67.0 (6.9) | 66.8 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 142 | 140 | 140 | 422
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 142 | 140 | 140 | 422
Region of Enrollment [Number; unit: participants]
  Japan | 142 | 140 | 140 | 422
Baseline (Visit 3) Benign Prostatic Hyperplasia Severity [Number; unit: participants] — Participants with BPH were defined as having had signs and symptoms of benign prostatic hyperplasia (BPH) (as diagnosed by a qualified physician) >6 months at Visit 1. Signs and symptoms of BPH included those associated with voiding (obstructive symptoms, such as incomplete emptying, intermittency, weak stream, straining)and/or storage (irritative symptoms, such as frequency, urgency, or nocturia).
  participants
    Moderate | 100 | 102 | 100 | 302
    Severe | 42 | 38 | 40 | 120
Current Alcohol Use [Number; unit: participants]
  Yes | 96 | 92 | 93 | 281
  No | 46 | 48 | 47 | 141
Current Tobacco Use [Number; unit: participants]
  Yes | 31 | 28 | 25 | 84
  No | 61 | 72 | 70 | 203
  Unknown or Not Recorded | 50 | 40 | 45 | 135
Previous Alpha-blocker Use [Number; unit: participants] — Actual use of alpha-blockers within the previous 12 months.
  participants
    Yes | 111 | 108 | 106 | 325
    No | 31 | 32 | 34 | 97
Previous Benign Prostatic Hyperplasia Therapy [Number; unit: participants] — Actual benign prostatic hyperplasia (BPH) therapy within the previous 12 months.
  participants
    Yes | 27 | 33 | 23 | 83
    No | 115 | 107 | 117 | 339
Previous Overactive Bladder Therapy [Number; unit: participants] — Actual overactive bladder (OAB) therapy within the previous 12 months.
  participants
    Yes | 10 | 12 | 7 | 29
    No | 132 | 128 | 133 | 393
Body Mass Index [Mean (Standard Deviation); unit: kilograms/meters squared] — Body mass index (BMI) is an estimate of body fat based on body weight divided by height squared.
  kilograms/meters squared | 23.3 (2.4) | 23.5 (2.6) | 23.6 (2.9) | 23.5 (2.6)
Duration of BPH [Mean (Standard Deviation); unit: years] — Participants had signs and symptoms of benign prostatic hyperplasia (BPH) (as diagnosed by a qualified physician) >6 months at Visit 1.
  years | 4.1 (3.0) | 4.5 (3.3) | 4.1 (2.9) | 4.2 (3.1)
Height [Mean (Standard Deviation); unit: centimeters] | 166.0 (5.9) | 166.9 (6.1) | 166.3 (6.3) | 166.4 (6.1)
Postvoid Residual Volume [Mean (Standard Deviation); unit: mililiters] — Postvoid residual volume (PVR) was measured by ultrasound at regular intervals.
  mililiters | 35.2 (46.6) | 32.2 (36.4) | 31.6 (42.7) | 33.0 (42.1)
Weight [Mean (Standard Deviation); unit: kilograms] | 64.4 (8.6) | 65.4 (8.3) | 65.4 (10.2) | 65.1 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) Total Score at 12-Week Endpoint
Description: The IPSS Total Score is obtained by combining the scores of the responses to 1 through 7 component questions. Each question is scored from 0-5 for an IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms.
Time Frame: Baseline, 12 weeks
Population: Participants in the Full Analysis Set (FAS): participants who were randomized and started study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 142 | 140 | 139
units on a scale | -4.5 (0.4) | -4.9 (0.4) | -3.8 (0.4)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.201, ANCOVA; With effects for treatment, prior alpha blocker use (yes/no), and baseline value; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.8 to 0.4], Standard Error of Mean 0.6 — Least Squares Mean Difference = Tadalafil 2.5 mg - Placebo
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p = 0.062, ANCOVA; With effects for treatment, prior alpha blocker use (yes/no) and baseline value; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.2 to 0.1], Standard Error of Mean 0.6 — Least Squares Mean Difference = Tadalafil 5 mg - Placebo

2. Secondary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) Storage (Irritative) Subscore at 12-Week Endpoint
Description: IPSS storage (irritative) subscore is the sum of Questions 2, 4 and 7 of the IPSS questionnaire. Scores range from 0 (not at all) to 5 (frequent irritative symptoms), thus the 3 questions of the irritative subscore range from 0 to 15.
Time Frame: Baseline, 12 weeks
Population: Participants in the Full Analysis Set (FAS): participants who were randomized and started study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 142 | 140 | 139
units on a scale | -1.6 (0.2) | -1.6 (0.2) | -1.4 (0.2)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.356, ANCOVA; With effects for treatment, prior alpha blocker use (yes/no) and baseline value; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.7 to 0.2], Standard Error of Mean 0.2 — Least Squares Mean Difference = Tadalafil 2.5 mg - Placebo
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p = 0.487, ANCOVA; With effects for treatment, prior alpha blocker use (yes/no) and baseline value; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.6 to 0.3], Standard Error of Mean 0.2 — Least Squares Mean Difference = Tadalafil 5 mg - Placebo

3. Secondary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) Voiding (Obstructive) Subscore at 12-Week Endpoint
Description: IPSS obstructive subscore is the sum of Questions 1, 3, 5 and 6 of the IPSS questionnaire. Scores range from 0 (not at all) to 5 (frequent obstructive symptoms), thus the 4 questions of the obstructive score range from 0 to 20.
Time Frame: Baseline, 12 weeks
Population: Participants in the Full Analysis Set (FAS): participants who were randomized and started study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 142 | 140 | 139
units on a scale | -2.9 (0.3) | -3.3 (0.3) | -2.4 (0.3)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.228, ANCOVA; With effects for treatment, prior alpha blocker use (yes/no) and baseline value; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.3 to 0.3], Standard Error of Mean 0.4 — Least Squares Mean Difference = Tadalafil 2.5 mg - Placebo
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p = 0.033, ANCOVA; With effects for treatment, prior alpha blocker use (yes/no) and baseline value; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.7 to -0.1], Standard Error of Mean 0.4 — Least Squares Mean Difference = Tadalafil 5 mg - Placebo

4. Secondary Outcome: Change From Baseline in IPSS Quality of Life (QoL) Index at 12-Week Endpoint
Description: Assessment of quality of life (QOL) by urinary symptoms, with scores ranging from 0 (delighted) to 6 (terrible).
Time Frame: Baseline, 12 weeks
Population: Participants in the Full Analysis Set (FAS): participants who were randomized and started study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 142 | 140 | 139
units on a scale | -0.5 (0.1) | -0.7 (0.1) | -0.4 (0.1)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.249, ANCOVA; With effects for treatment,BPH severity (moderate/severe), prior alpha blocker use (yes/no), and baseline value; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.1 — Least Squares Mean Difference = Tadalafil 2.5 mg - Placebo
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p = 0.022, ANCOVA; With effects for treatment,BPH severity (moderate/severe), prior alpha blocker use (yes/no) and baseline value; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to -0.0], Standard Error of Mean 0.1 — Least Squares Mean Difference = Tadalafil 5 mg - Placebo

5. Secondary Outcome: Change From Baseline in Overactive Bladder Symptom Score (OABSS) at 12-Week Endpoint
Description: The OABSS is a four-symptom questionnaire to assess overactive bladder (OAB) symptoms: daytime frequency, nighttime frequency, urgency, and urgency incontinence. Scores range from 0 - 15, with higher scores indicating more severe OAB symptoms.
Time Frame: Baseline, 12 weeks
Population: Participants in the Full Analysis Set (FAS): participants who were randomized and started study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 142 | 140 | 139
units on a scale | -0.7 (0.1) | -0.8 (0.1) | -0.7 (0.1)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.904, ANCOVA; with effects for treatment,BPH severity (moderate/severe), prior alpha blocker use (yes/no), and baseline value; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.4 to 0.3], Standard Error of Mean 0.2 — Least Squares Mean Difference = Tadalafil 2.5 mg - Placebo
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p = 0.800, ANCOVA; With effects for treatment, BPH severity(moderate/severe), prior alpha blocker use (yes/no), and baseline value; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.4 to 0.3], Standard Error of Mean 0.2

6. Secondary Outcome: Change From Baseline in Uroflowmetry Parameter: Peak Flow Rate (Qmax) at 12-Week Endpoint
Description: Uroflowmetry was assessed by Qmax, defined as the peak urine flow rate (measured in mL/second using a standard calibrated flowmeter).
Time Frame: Baseline, 12 weeks
Population: Participants in the Full Analysis Set (FAS): participants who were randomized and started study medication.
Measure: Least Squares Mean (Standard Error); unit: milliliters per second
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 140 | 135 | 136
milliliters per second | 0.7 (0.3) | 0.6 (0.3) | 1.4 (0.3)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.147, ANCOVA; With effects for treatment, BPH severity (moderate/severe), prior alpha blocker use (yes/no), and baseline value; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.5 to 0.2], Standard Error of Mean 0.4 — Least Squares Mean Difference = Tadalafil 2.5 mg - Placebo
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p = 0.094, ANCOVA; With effects for treatment, BPH severity (moderate/severe), prior alpha blocker use (yes/no), and baseline value; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.6 to 0.1], Standard Error of Mean 0.4 — Least Squares Mean Difference = Tadalafil 5 mg - Placebo

7. Secondary Outcome: Tadalafil Pharmacokinetics in Japanese Men: Plasma Concentration Measurement
Description: Plasma from participants in the tadalafil treatment groups were assayed using a validated liquid chromatographic/mass spectrometric (LC/MS) method.
Time Frame: Baseline, 12 weeks
Population: Participants who received 2.5 mg or 5 mg tadalafil once daily during the double-blind period.
Measure: Geometric Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg
Number analyzed (Participants) | 135 | 128
nanogram/milliliter
  0-6 hours (n=225, 200) | 86.0 (44.0) | 169 (41.2)
  6-12 hours (n=72, 72) | 68.7 (37.6) | 140 (51.3)
  12-24 hours (n=102, 106) | 57.5 (49.1) | 93.6 (55.6)
  24-48 hours (n=11, 8) | 43.5 (89.7) | 75.2 (56.0)

8. Secondary Outcome: Number of Participants With Adverse Events During 12 Weeks of the Study
Description: A listing of Adverse Events are reported in the Reported Adverse Event Section.
Time Frame: Baseline through 12 weeks
Population: All randomized participants
Measure: Number; unit: participants
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 142 | 140 | 140
participants
  Serious Adverse Events | 2 | 2 | 1
  Non-Serious Adverse Events | 52 | 54 | 53

9. Secondary Outcome: Change From Baseline in Blood Pressure at 12-Week Endpoint
Time Frame: Baseline, 12 weeks
Population: Safety Analysis Set: all randomized participants who received study treatment grouped by the treatment actually taken.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 142 | 140 | 139
mmHg
  Systolic Blood Pressure | -2.0 (11.9) | -3.4 (12.2) | -0.5 (14.0)
  Diastolic Blood Pressure | -0.7 (9.5) | -2.9 (8.3) | -0.9 (10.1)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.342, Wilcoxin rank-sum test — P-Value for systolic blood pressure
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p = 0.127, Wilcoxin rank sum test — P-Value for systolic blood pressure
Statistical Analysis 3: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.705, Wilcoxin rank-sum test — P-Value for diastolic blood pressure
Statistical Analysis 4: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p = 0.173, Wilcoxin rank-sum test — P-Value for diastolic blood pressure

10. Secondary Outcome: Change From Baseline in Sitting Heart Rate at 12-Week Endpoint
Time Frame: Baseline, 12 Weeks
Population: Safety Analysis Set: all randomized participants who received study treatment grouped by the treatment actually taken.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 142 | 140 | 139
beats per minute | -0.7 (9.9) | -1.2 (9.8) | 0.0 (8.2)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.606, Wilcoxin rank-sum test
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p = 0.149, Wilcoxin rank-sum test

11. Secondary Outcome: Change From Baseline in Postvoid Residual Volume (PVR) at 12-Week Endpoint
Description: Postvoid residual volume (PVR) is measured by ultrasound at regular intervals.
Time Frame: Baseline, 12 weeks
Population: Safety Analysis Set: all randomized participants who received study treatment grouped by the treatment actually taken.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 142 | 140 | 137
milliliters | -9.41 (41.43) | -5.15 (40.32) | -4.72 (36.40)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.428, Wilcoxin rank-sum test
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p = 0.426, Wilcoxin rank-sum test

12. Secondary Outcome: Change From Baseline in Prostate Specific Antigen (PSA) at 12-Week Endpoint
Description: Measurement of nanograms of PSA per milliliter (ng/mL) of blood.
Time Frame: Baseline, 12 weeks
Population: Safety Analysis Set: All randomized participants who received study treatment grouped by the treatment actually taken.
Measure: Mean (Standard Deviation); unit: Micrograms per liter
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 142 | 138 | 139
Micrograms per liter | 0.26 (1.54) | 0.09 (0.88) | 0.14 (2.90)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.060, Wilcoxin rank-sum
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p = 0.212, Wilcoxin rank-sum

13. Secondary Outcome: Change From Baseline in the International Prostate Symptom Score (IPSS) Total Score at 54-Week Endpoint
Description: as for outcome 1
Time Frame: Baseline, 54 weeks
Population: All participants enrolled in the open-label extension period who received at least 1 dose of tadalafil.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 135 | 128 | 131
units on a scale | -5.2 (5.9) | -5.4 (6.3) | -6.2 (5.4)

14. Secondary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) Storage (Irritative) Subscore at 54-Week Endpoint
Description: as for outcome 2
Time Frame: Baseline, 54 weeks
Population: All participants enrolled in the open-label extension period who received at least 1 dose of tadalafil.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 135 | 128 | 131
units on a scale | -1.9 (2.5) | -1.6 (2.8) | -1.8 (2.5)

15. Secondary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) Voiding (Obstructive) Subscore at 54-Week Endpoint
Description: as for outcome 3
Time Frame: Baseline, 54 weeks
Population: All participants enrolled in the open-label phase who received at least 1 dose of tadalafil.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 135 | 128 | 131
units on a scale | -3.4 (4.1) | -3.7 (4.5) | -4.3 (3.9)

16. Secondary Outcome: Change From Baseline in IPSS Quality of Life (QoL) Index at 54-Week Endpoint
Description: Assessment of quality of life (QOL) by urinary symptoms, with scores ranging from 0 (delighted) to 6 (terrible).
Time Frame: Baseline, 54 weeks
Population: All participants enrolled in the open-label extension who received at least 1 dose of tadalafil.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 135 | 128 | 131
units on a scale | -0.8 (1.2) | -1.0 (1.4) | -0.9 (1.4)

17. Secondary Outcome: Change From Baseline in Overactive Bladder Symptom Score (OABSS) at 54-Week Endpoint
Description: as for outcome 5
Time Frame: Baseline, 54 weeks
Population: All participants enrolled in the open-label extension who received at least 1 dose of tadalafil.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 135 | 128 | 131
units on a scale | -0.9 (2.0) | -1.0 (2.4) | -0.9 (2.0)

18. Secondary Outcome: Change From Baseline in Uroflowmetry Parameter: Peak Flow Rate (Qmax) at 54-Week Endpoint
Description: as for outcome 6
Time Frame: Baseline, 54 weeks
Population: All participants enrolled in the open-label extension who received at least 1 dose of tadalafil.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 134 | 128 | 127
units on a scale | 2.29 (4.29) | 1.51 (4.48) | 2.01 (5.05)

19. Secondary Outcome: Number of Participants With Adverse Events During 42 Weeks of Open-Label Treatment
Description: A listing of Adverse Events are reported in the Reported Adverse Event Section.
Time Frame: End of 12 weeks of double-blind through 54 weeks
Population: All participants enrolled in the open-label extension who received at least 1 dose of tadalafil.
Measure: Number; unit: participants
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 135 | 128 | 131
participants
  Serious Adverse Events | 3 | 4 | 4
  Non-Serious Adverse Events | 81 | 81 | 94

20. Secondary Outcome: Change From Baseline in Blood Pressure During at 54-Week Endpoint
Time Frame: Baseline, 54 weeks
Population: All participants enrolled in the open-label extension who received at least 1 dose of tadalafil.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 135 | 128 | 131
millimeters of mercury (mmHg)
  Systolic blood pressure | -2.1 (13.4) | -1.2 (13.2) | -0.5 (14.2)
  Diastolic blood pressure | -1.6 (9.6) | -2.9 (9.2) | -1.3 (9.8)

21. Secondary Outcome: Change From Baseline in Sitting Heart Rate at 54-Week Endpoint
Time Frame: Baseline, 54-weeks
Population: All participants enrolled in the open-label extension who received at least 1 dose of tadalafil.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 135 | 128 | 131
beats per minute (bpm) | 1.4 (10.4) | 0.4 (9.3) | 2.1 (10.6)

22. Secondary Outcome: Change From Baseline in Prostate Specific Antigen (PSA) at 54-Week Endpoint
Description: Measurement of nanograms of PSA per milliliter (ng/mL) of blood.
Time Frame: Baseline, 54 weeks
Population: All participants enrolled in the open-label extension who received at least 1 dose of tadalafil.
Measure: Mean (Standard Deviation); unit: microgram/liter
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 135 | 127 | 129
microgram/liter | 0.4 (1.0) | 0.3 (0.9) | 0.3 (1.4)

23. Secondary Outcome: Change From Baseline in Postvoid Residual Volume (PVR) at 54-Week Endpoint
Description: Post residual volume (PVR) is measured by ultrasound at regular intervals.
Time Frame: Baseline, 54 weeks
Population: All participants enrolled in the open-label extension who received at least 1 dose of tadalafil.
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 135 | 128 | 131
milliliter | -5.7 (50.0) | -1.9 (42.9) | -5.5 (46.8)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) - defined as events that 1st occurred/worsened after randomization at Week 0.
Description: Post-baseline period began after enrollment (Week 12) in open-label extension. If subject reports the occurrence of an event more than once, the most severe of those events was used to determine if event was TE. Analysis of TEAEs was summarized for open-label extension alone (Weeks 12-54). Week 0 of double-blind treatment period was baseline.
Groups:
- Tadalafil 2.5 mg - Double-Blind Phase: 2.5 milligrams (mg) tadalafil tablet by mouth once a day for 12 weeks followed by 5 mg tadalafil tablet by mouth once a day for 42 weeks in the Open-Label Phase.
- Tadalafil 5 mg - Double-Blind Phase: 5 mg tadalafil tablet by mouth once a day for 12 weeks then continue 5 mg tadalafil tablet by mouth once a day for 42 weeks during the Open-Label Phase.
- Placebo - Double-Blind Phase: Placebo tablet taken by mouth once a day for 12 weeks.
  Then subjects may take 5 mg tadalafil tablet by mouth once a day for 42 weeks during the Open-Label Phase.
- Tadalafil 2.5 mg: Tadalafil 5 mg Open-Label: 5 mg tadalafil tablet by mouth once a day for 42 weeks. Participants had previously received 2.5 mg tadalafil in the double-blind phase.
- Tadalafil 5 mg: Tadalafil 5 mg Open-Label: 5 mg tadalafil tablet by mouth once a day for 42 weeks. Participants had previously received 5 mg tadalafil in the double-blind phase.
- Placebo: Tadalafil 5 mg Open-Label: 5 mg tadalafil tablet by mouth once a day for 42 weeks. Participants had previously received placebo in the double-blind phase.
Arm/Group | Tadalafil 2.5 mg - Double-Blind Phase | Tadalafil 5 mg - Double-Blind Phase | Placebo - Double-Blind Phase | Tadalafil 2.5 mg: Tadalafil 5 mg Open-Label | Tadalafil 5 mg: Tadalafil 5 mg Open-Label | Placebo: Tadalafil 5 mg Open-Label
Serious Adverse Events (participants affected / at risk) | 2/142 | 2/140 | 1/140 | 3/135 | 4/128 | 4/131
Other Adverse Events (participants affected / at risk) | 52/142 | 54/140 | 53/140 | 81/135 | 81/128 | 94/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil 2.5 mg - Double-Blind Phase (N=142) | Tadalafil 5 mg - Double-Blind Phase (N=140) | Placebo - Double-Blind Phase (N=140) | Tadalafil 2.5 mg: Tadalafil 5 mg Open-Label (N=135) | Tadalafil 5 mg: Tadalafil 5 mg Open-Label (N=128) | Placebo: Tadalafil 5 mg Open-Label (N=131)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil 2.5 mg - Double-Blind Phase (N=142) | Tadalafil 5 mg - Double-Blind Phase (N=140) | Placebo - Double-Blind Phase (N=140) | Tadalafil 2.5 mg: Tadalafil 5 mg Open-Label (N=135) | Tadalafil 5 mg: Tadalafil 5 mg Open-Label (N=128) | Placebo: Tadalafil 5 mg Open-Label (N=131)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 3 (3) | 0 (0) | 4 (4) | 3 (3) | 2 (2)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 5 (5) | 8 (16) | 11 (12) | 12 (13)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) | 4 (4) | 6 (7) | 5 (6)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 5 (5) | 2 (2) | 3 (3)
Gastritis atrophic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periproctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reflux oesophagitis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 5 (5) | 4 (4) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 5 (5)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (11) | 14 (14) | 18 (19) | 25 (28) | 15 (17) | 19 (31)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (5)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour marker increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 7 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 2 (2) | 5 (5) | 5 (5) | 8 (8)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 3 (3) | 9 (9)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nipple disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (4) | 3 (4) | 6 (6)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental implantation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal tube insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Internal fixation of fracture (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Ureteral catheterisation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (3) | 2 (2) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 4 (4) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days